CLINICAL TRIAL: NCT04446702
Title: Retrospective Real-life Study From One Brazilian Reference Centre Assessing Long-term Experience in the Treatment of Adult Spasticity With AbobotulinumtoxinA (RETURN Study)
Brief Title: Retrospective Real-Life Study From One Brazilian Reference Center Assessing Long-Term Experience In The Treatment Of Adult Spasticity With AbobotulinumtoxinA
Acronym: RETURN
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-BR-52120-269
Record Dates: First submitted 2020-06-08; First posted 2020-06-25 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe the long-term use of abobotulinumtoxinA (Dysport®) in adult subjects affected with upper limb spasticity (ULS) +/- lower limb spasticity (LLS) who received treatment with Dysport® for a minimum of three injections cycles at the Instituto de Medicina Física e Reabilitação do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (IMREA HC FMUSP) in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥18 years old at the time of the first Dysport® injection
* Diagnosed with spasticity
* Treated with a minimum of three Dysport® injection cycles for ULS +/- LLS in the observational period
* Follow up effectiveness data are available in the subject's medical record

Exclusion Criteria:

* Patients have received previous treatment with another BoNT-A less than 12 weeks prior to the patient data collection in the study
* Adults with cerebral palsy
* Patients treated with BoNT-A in a clinical trial setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible adult patients having received Dysport® for at least three cycles for the treatment of ULS +/- LLS between January 1st, 2006 and July 31st, 2019 at Instituto de Medicina Física e Reabilitação do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (IMREA HC FMUSP) in Brazil with pre- and post-injection effectiveness data available will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Average total dose injected during all sessions of Dysport® in ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Median total dose injected during all sessions of Dysport® in ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Average interval between Dysport® injections in ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)

SECONDARY OUTCOMES:
Baseline subjects characteristics | Baseline (first Dysport® injection)
  * Demography (age at first injection during the period of interest, sex, weight)
  * History of spasticity
Total number of Dysport® injection cycles | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Total time exposure to Dysport® treatment in ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Total dose injected per cycle, per limb, per muscle and overall | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Number of muscles injected in ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Reported reason for Dysport® injection and for change | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  Outcome will be assessed according following reasons: due to medical need, unplanned need and not recorded
Number of Dysport® interruptions | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
Reasons of Dysport® discontinuation | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019).
  Outcome will be assessed according following reasons: side effects (e.g. excessive weakness, hematoma), contractures, absence of clinical response, long lasting clinical improvement, patient lost follow up and other.
Changes in Modified Ashworth Scale (MAS) scores by time period per muscle | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  The MAS is a six-point scale to grade muscle tone in the injected muscle from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension). Upper limb: shoulder abduction, elbow flexion, elbow extension, wrist flexion, wrist extension and fingers flexion. Lower limb: hip flexion, hip adduction, hip abduction, knee flexion, knee extension, ankle dorsiflexion and ankle plantar flexion.
Changes in Functional Independence Measure (FIM) subscales | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  Subscales and total scores of FIM will be measured. The FIM is a method for categorising patients on a seven-point scale (range 1 to 7). It comprises of 18 items, grouped into 2 subscales (motor and cognition). The motor subscale includes: eating, grooming, bathing, dressing upper body, dressing lower body, toileting, bladder management, bowel management, transfers - bed/chair/wheelchair, transfers - toilet, transfers - bath/shower, walk/wheelchair and stairs. The cognition subscale includes: comprehension, expression, social interaction, problem solving and memory. The Scores are summed to obtain a total score that can range between 18 and 126.
Changes in Pain score according to pain Visual Analogue Scales (VAS) | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  The pain Visual Analogue Scale (VAS) is a numeric graphic rating scale (NGRS) of self-reported symptoms. Scores are recorded as whole numbers between zero and 10, where zero indicates no pain symptom at all, and 10 indicates a as bad as it could be.
Gait pattern evaluation in patients with LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  Gait Pattern Modification in patients with LLS is based on physician´s clinical evaluation and it will be evaluated for each lower limb (left and right) or both according to pre-specified patterns: equinismus, foot inversion, knee hyperextension, adduction, mowing abduction, thigh elevation, hip elevation, false trendelenburg, not able to walk. The Gait Pattern Improvement is described based on patient´s perception of gait. The patients respond Yes or No and if Yes the % of improvement is replied
Concomitant drugs for the management of patients with ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  List the systemic drug therapies, including: antispasticity medications (e.g. Baclofen, Tizanidin, Dantrolene), simple pain medications (e.g. paracetamol or NSAIDS), neuropathic pain and spasticity medications (e.g. Gabapentin, Pregabalin, Amitriptyline), opioids, phenol, alcool or other neurolytic agents.
Non-drug concomitant therapies for the management of patients with ULS +/- LLS | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  List the non-drug concomitant therapies, including occupational therapy, physiotherapy and others (e.g.: orthotics, serial casting, splinting, electric stimulation)
Incidence and intensity of Adverse Events | From baseline (visit 1) and up to the last injection during data record (January 1st, 2006 to July 31st, 2019)
  Adverse events will be assessed according to incidence, intensity/grade (mild, moderate and severe), causality (related and not related to the product), outcome (the overall association between an exposure to a drug and an outcome) and action taken. All Adverse Events (AEs) (including fatal events and Serious Adverse Events (SAEs)) and special situation (pregnancy, overdose, off-label use) will be reported with the number and proportion of events. The incidence will be provided and classified by System Organ Class and Preferred Term

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Instituto de Medicina Física e Reabilitação do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (IMREA HC FMUSP), São Paulo, Brazil